CLINICAL TRIAL: NCT04721366
Title: Gaucher Disease During Infancy and Early Childhood and Experience With Enzyme Replacement Therapy (ERT) Using Velaglucerase Alfa (VPRIV): A Combined Retrospective and Prospective Cohort Study
Brief Title: A Study of Velaglucerase Alfa (VPRIV) Given as Standard Patient Care in Young Children With Gaucher Disease
Acronym: PEDS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MACS-2020-052801; TAK-669-4019 (Other: Takeda)
Record Dates: First submitted 2021-01-21; First posted 2021-01-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care (SoC): Neonatal and pediatric participants who has been on ERT (VPRIV) will be followed up for 36 months from the time of treatment initiation as per SOC.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Neonatal and pediatric participants who has been on ERT (VPRIV) will be assessed as per SOC.
  Other Names: SOC

SUMMARY:
The main aim of this study is to learn if velaglucerase alfa (VPRIV) improves growth and symptoms in participants up to 5 years of age with Gaucher disease. Symptoms will be checked with blood tests.

This study is about collecting data available in the participant's medical record as well as data from each participant's ongoing treatment. No study medicines will be provided to participants in this study. The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

When the participants start the study, they will visit the study clinic every 6 months after their first visit.

ELIGIBILITY:
Inclusion Criteria:

* The participant's caregiver is able and willing to provide informed consent.
* The participant is male or female younger than or equal to 4 years of age at treatment initiation.
* The participant has received and confirmed a current diagnosis of GD type 1 or type 3 (biochemically and/or genetically).
* The participant has been receiving intravenous (IV) Velaglucerase alfa treatment for GD.
* In the opinion of the investigator, the participant's caregiver is capable of understanding and complying with protocol requirements.
* The participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

* The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., child, sibling) or may consent under duress.
* The participant is judged by the investigator as being ineligible for any other reason.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal and pediatric participants included have a diagnosis of GD type I and III and are currently being treated with total ERT (VPRIV) for less than or equal to (<=) 36 months from the time of treatment initiation.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin (Hb) Level | From start of ERT initiation up to 5 years of age
  Increase hemoglobin levels up to 11.0 gram per deciliter (g/dL) will be assessed.
Percent Change From Baseline in Platelet Count Increase | From start of ERT initiation up to 5 years of age
  Percent change from baseline for platelet count increase will be assessed.
Percent Change From Baseline in Liver Volume | From start of ERT initiation up to 5 years of age
  Percent change from baseline in liver volume will be assessed.
Percent Change From Baseline for Spleen Volume | From start of ERT initiation up to 5 years of age
  Percent change from baseline for spleen volume will be assessed.
Percentage of Participants With Growth Normalization | From start of ERT initiation up to 5 years of age
  Percentage of participants with growth normalization will be assessed.
Percentage of Participants With Improvement in Bone Disease | From start of ERT initiation up to 5 years of age
  Percentage of participants with improvement in bone disease will be assessed.
Percentage of Participants With Improvement in Thrombocytopenia | From start of ERT initiation up to 5 years of age
  Percentage of participants with improvement in thrombocytopenia will be assessed.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From start of ERT initiation up to 5 years of age
  An adverse event (AE) is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An SAE is any event that results in: death; life-threatening; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly/birth defect or a medically important event. AEs include SAEs, non-serious AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Lysosomal & Rare Disorders Research & Treatment Center, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/600e8bb0565ce300294c6ae8